CLINICAL TRIAL: NCT05654727
Title: Cognitive Impairment and BDNF in Patients With Diabetes and Prediabetes
Brief Title: Cognitive Functions and BDNF in T2DM and Prediabetes Patients
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: bsekerci1
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Type 2; PreDiabetes; Cognitive Impairment
Keywords: diabetes; BDNF; T2DM; prediabetes; cognition
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Cognitive Dysfunction; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type 2 Diabetes Mellitus
- Prediabetes
- Healthy Control

SUMMARY:
Clinical and epidemiological studies suggest links between cognitive impairments and Type 2 diabetes (T2DM). The underlying mechanisms and causality in diabetes-related cognitive impairment are largely unknown. The aim of this study is to investigate cognitive impairment and the role of BDNF in prediabetes and diabetes patients.

DETAILED DESCRIPTION:
Cognitive dysfunction is increasingly recognized as a common complication and comorbidity in both type 1 and type 2 diabetes (T2DM). Due to the increasing incidence of diabetes and the life expectancy of individuals with T2DM, it is important to determine the cognitive problems and related factors in these patients. Cognitive impairment can be observed in all age groups in individuals with diabetes, and its severity can range from mild cognitive impairment to dementia. Although there are few studies in the literature investigating cognitive impairment in prediabetes, it is not clear whether it is a risk factor.

The number of studies investigating biomarkers of potential importance for understanding changes in the brain of T2DM patients is increasing rapidly. The relationship of biomarkers associated with the main pathologies of dementia, including Alzheimer's disease (AD) and vascular disease, as well as various biomarkers associated with brain parenchymal damage, blood flow and metabolism, with the cognitive status of diabetic patients are investigated. It has been determined in animal experiments that Brain Induced Neurotrophic Factor (BDNF) may be among the molecular factors linking T2DM with dementia neuropathology. It has also been stated that high glucose levels are associated with cognitive impairment and total hippocampal volume reductions, and hippocampal changes can be used as an early marker of diabetes-related brain damage. Considering that the expression of BDNF in the brain is high in hippocampus neurons, it may be an early marker of cognitive impairment in diabetes.

This research is a cross-sectional observational study. The aim of this study is to investigate cognitive impairment and the role of BDNF in prediabetes and diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* age from 30 to 65 years
* having at least primary school education

Exclusion Criteria:

* severe psychiatric (e.g,major depressive disorder) or neurologic disorder (demyelinating diseases, stroke or brain tumor)
* using insulin (Insulin therapy was taken as an exclusion criterion to avoid the effect of hypoglycemia on cognition)
* vision and hearing problem
* Hypothyroidism, B12 and folic acid deficiency
* Advanced chronic renal failure (stage 4-5)
* uncontrolled hypertension
* patients with hypoglycemia-hyperglycemia attacks
* Alcohol, substance addiction.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetes, prediabetes and control patients who applied to the internal medicine outpatient clinic of Bezmialem Vakıf University and met the inclusion/exclusion conditions of the study
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Cognitive Functions | baseline
  MoCA total score and subscores were used to evalaute cognitive functions
BDNF | baseline
  Serum BDNF were evaluated by Elisa

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)